CLINICAL TRIAL: NCT01727154
Title: Immune Monitoring Protocol in Men With Prostate Cancer Enrolled in a Clinical Trial of Sipuleucel-T
Acronym: PRIME
Status: Terminated | Type: Observational
Why Stopped: Administrative reasons
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Other Study IDs: P11-4
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, manufacturing samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sipuleucel-T
  Interventions: Biological: Sipuleucel-T

INTERVENTIONS:
Biological: Sipuleucel-T — Each dose of sipuleucel-T contains a minimum of 50 million autologous CD54+ cells activated with PAP-GM-CSF. The recommended course of therapy for sipuleucel-T is 3 complete doses, given at approximately 2-week intervals.
  Other Names: PROVENGE; APC8015

SUMMARY:
The purpose of this study is to evaluate the immune response induced by sipuleucel-T (Provenge®).

DETAILED DESCRIPTION:
Subjects will receive sipuleucel-T, and potentially other medications, as part of the clinical trial in which they are concurrently enrolled. For this study, cellular and humoral immune responses will be assessed. No additional study treatments will be conducted beyond what is required for the subject's concurrent clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Subjects with prostate cancer who are enrolled in a clinical trial of sipuleucel-T (including a Dendreon-sponsored clinical trial or registry, or an IIT)
* Subjects have not yet undergone leukapheresis for their first dose of sipuleucel-T
* Subjects must understand and sign an informed consent form prior to their first leukapheresis

Exclusion Criteria:

•None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men at least 18 years of age with prostate cancer who are enrolled in a clinical trial of sipuleucel-T (including a Dendreon-sponsored clinical trial or registry, or an IIT), and have not yet undergone leukapheresis for their first dose of sipuleucel-T.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2012-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Brown, MD, Study Director — Dendreon Pharmaceuticals, LLC
Locations (39):
- United States (39):
  - 21st Century Oncology, Scottsdale, Arizona
  - Tower Urology / Tower Research Institute, Los Angeles, California
  - Prostate Oncology Specialists, Inc., Marina del Rey, California
  - The Urology Center of Colorado, Denver, Colorado
  - Howard University Cancer Center, Washington D.C., District of Columbia
  - First Urology, PSC, Jeffersonville, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Tulane University, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - St. Louis Cancer Care, LLP, Bridgeton, Missouri
  - St. Louis Cancer Care, LLP, St Louis, Missouri
  - Southeast Nebraska Hematology & Oncology Consultants, P.C. d/b/a Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Delaware Valley Urology, LLC, Mount Laurel, New Jersey
  - National Translational Research Group, Inc., East Setauket, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Urology Partners, Gastonia, North Carolina
  - Raleigh Hematology Oncology Associates, D.B.A., Cancer Centers of North Carolina, Raleigh, North Carolina
  - TriState Urologic Services PSC Inc., dba The Urology Group, Cincinnati, Ohio
  - Urologic Specialists of Oklahoma, Tulsa, Oklahoma
  - Providence Health & Services, Portland, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Northwest Cancer Specialists, PC, Tualatin, Oregon
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Centerl, Seattle, Washington
  - Northwest Cancer Specialists, Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sipuleucel-T
Started | 139
Completed | 80
Not Completed | 59
Not completed — Death | 17
Not completed — Withdrawal by Subject | 14
Not completed — Subject Withdrew Consent | 18
Not completed — Study Terminated | 6
Not completed — No Discontinuation Documentation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 115
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 139
Height [Mean (Standard Deviation); unit: Centemeters] | 177.6 (6.8)
Weight [Mean (Standard Deviation); unit: Kg] | 91.1 (19.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (5.6)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour;3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair;5=Dead
  Participants
    ECOG=0 | 89
    ECOG=1 | 34
    ECOG=2 | 4
    ECOG=3 | 3
    Missing | 9
Gleason Sum Reported [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleson Sum<= 6 | 14
    Gleson Sum=7 | 37
    Gleson Sum>= 8 | 63
    Missing | 25

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Exhibit Any Immune Response at Any Post-treatment Time Point (6, 10, 14, 26, 39, and 52 Weeks After the First Infusion of Sipuleucel-T).
Description: The primary immune response analysis population will include all subjects who receive all 3 infusions of sipuleucel-T. The primary analysis will measure the percentage of subjects who exhibit any immune response at any post-treatment time point (6, 10, 14, 26, 39, and 52 weeks after the first infusion of sipuleucel-T).
Time Frame: Each subjects was to be followed for approximately 52 weeks beginning with the date of the subject's first infusion of siupleucel-T.
Population: This study was terminated early due to administrative reasons. A min of 200 patients were needed to obtain reliable data but only 139 were enrolled, 123 treated only 118 had analyzable immune response samples. Therefore this was a descriptive analysis of only 118pts with an immune response after dosing with Provenge. No comparative group available.
Measure: Count of Participants; unit: Participants
Arm/Group | Sipuleucel-T
Number analyzed (Participants) | 118
Participants
  Subjects who had an immune response | 110
  Subjects who did not have an immune response | 8

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not monitored/assessed. Reporting requirements for serious adverse events (SAEs) are described in the respective protocols (P10-3 and P12-1) for the trial in which each subject is concurrently enrolled.
Description: All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
  Reporting requirements for serious adverse events (SAEs) are described in the respective protocols (P10-3 and P12-1) for the trial in which each subject is concurrently enrolled.
Arm/Group | Sipuleucel-T
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed as a minimum of 200 patients were needed to obtain reliable data; however only 123 were treated. Given the small number of patients enrolled, analyses do not provide reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT01727154/Prot_SAP_000.pdf